CLINICAL TRIAL: NCT00530140
Title: Idiotypic Vaccination for Poor-prognosis Follicular Lymphoma Patients in First Relapse
Brief Title: Idiotypic Vaccination for Follicular Lymphoma Patients
Acronym: FLIDVAX2006
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: University of Navarrra Hospital (Clinica Universitaria) (Other); Center for Applied Medical Research (Centro de Investigación Médica Aplicada) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUN-90-2006
Record Dates: First submitted 2007-09-12; First posted 2007-09-17 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Follicular Lymphoma; First Relapse/Progression
Keywords: Follicular Lymphoma; Idiotype vaccine
MeSH Terms: conditions — Lymphoma, Follicular; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): All patients will receive the same vaccination schedule/formulation
  Interventions: Biological: Follicular lymphoma, patient-specific, soluble protein idiotype vaccine

INTERVENTIONS:
Biological: Follicular lymphoma, patient-specific, soluble protein idiotype vaccine — 0.5 mg of idiotype conjugated to 0.5 mg of KLH + 125 mcg of GM-CSF 5 monthly vaccinations followed by 3 bi-monthly vaccinations, followed by one boost every three months until either relapse or death from cause unrelated to lymphoma

SUMMARY:
Poor prognosis follicular lymphoma patients have an estimated median overall survival of 5-6 years. The proposed trial offers life-time idiotypic vaccination to all such patients in first relapse/progression who will achieve second (first, in the case of patients who have never achieved complete response following standard first-line treatment) complete response through autologous stem cell transplant prior to vaccination start. The ultimate goal is a cure, defined as a vaccine-maintained complete response lasting both at least 10 years and at least twice as long as each patient's first complete response.

DETAILED DESCRIPTION:
Idiotypic vaccination has already proved capable (in responding patients) of: biological efficacy, that is the capacity of inducing an idiotype- and tumor-specific immune response (Kwak LW et al. NEJM 1992); clinical efficacy, that is the capacity of inducing specific immune responses able to kill in vivo follicular lymphoma cells that had survived pre-vaccine chemotherapy (Bendandi M et al. Nature Med 1999): clinical benefit, that is the capacity of prolonging survival of responding patients (Inoges et al. JNCI 2006). Now, we want to test whether it is also capable of contributing to the ultimate goal of preventing relapse indefinitely in responding patients.

ELIGIBILITY:
Inclusion Criteria: at least one of the following:

* FLIPI score 3 thru 5 at diagnosis and/or at relapse
* First complete response shorter than 3 years, if no maintenance (Interferon, Rituximab, etc) treatment was administered, or than 5 years if maintenance treatment was administered
* No treatment has been able to induce complete response until autologous stem cell transplant
* Poor-prognosis genomic profiling

Exclusion Criteria: any of the following:

* Unavailability of a harvestable lymph node of at least cm 2x2x2
* Life expectancy < 1 year
* Abnormal heart or liver or kidney function
* ECOG Performance Status > 2
* Failure to sign informed consent before enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Primary Completion 2013-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who both never relapse and have a second complete response longer than their first response (cured) | 15 years

SECONDARY OUTCOMES:
Percentage of patients who successfully maintain a measurable, specific immune response throughout the active vaccination time frame | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: MAURIZIO BENDANDI, MD, PhD, Principal Investigator — University of Navarra
Locations (1):
- University of Navarra Hospital, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Inoges S, Rodriguez-Calvillo M, Zabalegui N, Lopez-Diaz de Cerio A, Villanueva H, Soria E, Suarez L, Rodriguez-Caballero A, Pastor F, Garcia-Munoz R, Panizo C, Perez-Calvo J, Melero I, Rocha E, Orfao A, Bendandi M; Grupo Espanol de Linfomas/Trasplante Autologo de Medula Oseo study group; Programa para el Estudio y Tratamiento de Hemopatias Malignas study group. Clinical benefit associated with idiotypic vaccination in patients with follicular lymphoma. J Natl Cancer Inst. 2006 Sep 20;98(18):1292-301. doi: 10.1093/jnci/djj358. PMID 16985248